CLINICAL TRIAL: NCT04095312
Title: A Prospective, Single-center, Single-group Clinical Study for Evaluating the Clinical Safety and Effectiveness of the Automated Robotic Robot, Revo-i Surgical Robot System (Model MSR-5100), Used for General Endoscopic Surgery.
Brief Title: Clinical Study for Evaluating the Clinical Safety and Effectiveness of the Automated Robotic Robot, Revo-i Surgical Robot System (Model MSR-5100), Used for General Endoscopic Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2019-0030
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Periampullary Cancer

STUDY DESIGN:
Intervention Model Description: In a study involving relatively small groups of 10 to 50 people, the study showed a high success rate of more than 90% similar to the study of more than 100 large groups, and the stability was well proven.
  total 33 patients (10 pancreaticobiliary tracts, 13 urinary tract areas, 10 colonic areas), the minimum number of clinical studies that can be statistically analyzed within the limits to meet the study objective of evaluating the "accuracy of procedure"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pancreaticobiliary disease (Experimental): 10 pancreaticobiliary disease cases
  Interventions: Procedure: Revo-i robotic surgery system (Model MSR-5100)
- Urinary tract disease (Experimental): 13 urinary tract disease cases
  Interventions: Procedure: Revo-i robotic surgery system (Model MSR-5100)
- Colon disease (Experimental): 10 colon disease cases
  Interventions: Procedure: Revo-i robotic surgery system (Model MSR-5100)

INTERVENTIONS:
Procedure: Revo-i robotic surgery system (Model MSR-5100) — for evaluating the clinical safety and effectiveness of the automated robotic robot, Revo-i Surgical Robot System (Model MSR-5100), used for general HBP surgery
  Other Names: Revo-I robotic surgery, davinci, pancreas cancer
  Arms: pancreaticobiliary disease
Procedure: Revo-i robotic surgery system (Model MSR-5100) — for evaluating the clinical safety and effectiveness of the automated robotic robot, Revo-i Surgical Robot System (Model MSR-5100), used for general Uro surgery
  Other Names: Revo-I robotic surgery, davinci, Urology
  Arms: Urinary tract disease
Procedure: Revo-i robotic surgery system (Model MSR-5100) — for evaluating the clinical safety and effectiveness of the automated robotic robot, Revo-i Surgical Robot System (Model MSR-5100), used for general colorectal surgery
  Other Names: Revo-I robotic surgery, davinci, colorectal cancer
  Arms: Colon disease

SUMMARY:
This study is based on the ergonomic features of the most common surgical procedures, which require advanced techniques and relatively difficult operations, such as pancreatobiliary surgery, prostatectomy, nephrectomy, colon and rectal resection. This study id designed to verify the clinical safety and effectiveness of 'Revo-i Surgical Robot System (Model MSR-5100), developed by Mirae Company to overcome the limitations of general laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

All of the following selection criteria must be met to be enrolled in this clinical trial.

* Common Standard

  1. Adults over 19
  2. Voluntary consent to clinical research and willingness to comply with the protocol
* Pancreaticobiliary tract area surgery

  1. A person deemed to need surgery for pancreaticobiliary tract due to one or more of the following reasons:

     * Benign and borderline periampullary cancer
     * Resectable masses (biliary cancer, pancreatic cancer, duodenal cancer, AoV cancer, etc.) Congenital gallbladder cysts
     * Endoscopic treatment of adenocarcinoma and early stage lesions of ampulla
     * There is no major organ or vascular invasion
     * Lack of severe pancreatitis and cholangitis
  2. Patients considering laparoscopic surgery who cannot perform da Vinci robot surgery due to personal expense
  3. Others who have been diagnosed with high latitude pancreaticobiliary tract surgery according to the researcher's judgment
* Prostatectomy

  1. Persons deemed necessary for prostatectomy in the following cases:

     -The prostate is at low risk or medium risk, and the tumor is located at the local site without metastasis Criteria for Prostate Risk Group Prostate low risk group Prostate Cancer Stage (T1-T2a) and Gleason Grade ≤6 and PSA <10ng / ml Risk group in the prostate Prostate cancer stage (T2b-T2c) or Gleason grade 7 or10 ng / ml ≤ PSA ≤ 20 ng / ml

     * Reference) NCCN (National Comprehensive Cancer Network), 2015
  2. Others who have been diagnosed as requiring prostate surgery according to the researcher's judgment
* Nephrectomy

  1. Persons deemed necessary for renal resection should:

     Localized renal cell carcinoma without metastasis to organs other than the kidney Stage 1A, IB, II, III

     * Reference) NCCN (National Comprehensive Cancer Network), 2011
  2. Others who have been diagnosed with nephrectomy according to the researcher's judgment
* Colon and Rectal Surgery

  1. A person who needs to have a resection for colon and rectal cancer

     * Histopathologically confirmed by adenocarcinoma of the rectum or colon
     * No remote transition (M0)
     * Primary tumor without other peripheral organ involvement (T1-T4a)
     * When intestinal obstruction is not accompanied In case of elective surgery
     * Does not require resection of any organ other than the primary tumor
  2. Others who have been diagnosed as having to need colon and rectal resection according to the researcher's judgment

Exclusion Criteria:

* Common Standard

  1. If you have mental illness or serious systemic disease
  2. Body Mass Index (BMI) ≥ 30, high obesity
  3. General anesthesia is not possible due to uncontrolled bleeding tendency or lowering of cardiopulmonary function
  4. If you have a positive or reactive pregnancy
  5. Patients who wish to undergo conventional laparoscopy or da Vinci robotic surgery
* Pancreaticobiliary tract area surgery

  -If you have a history of open abdominal surgery Liver cirrhosis Patients with abnormally inoperable pancreatobiliary malformations, other pancreatic biliary diseases, or systemic diseases
* Prostatectomy

  1. Surgical removal of prostate tumor is difficult or life expectancy is short
  2. Meets the exclusion criteria of prostatectomy below <Exclusion Criteria for Prostatectomy>

     * Clinical study subjects at high risk group Criteria of Prostate Risk Group Prostate High Risk Group Prostate Cancer Stage (T3a and above) or Gleason class ≥ 8 or ≤ 10 or PSA> 20ng / ml

       * Reference) NCCN (National Comprehensive Cancer Network), 2015
     * Have a history of surgery on the prostate, urethra, or bladder neck
     * If you have a history of open surgery
* Nephrectomy

  1. If you have a history of epigastric open surgery or have had kidney surgery
  2. History of chronic inflammation in the kidneys and the posterior cavity

  2) prone to bleeding 3) When a disease such as kidney or vascular malformation is impossible to the extent that surgery is impossible
* Colon and Rectal Surgery

  1. If you have a history of lower abdominal and pelvic laparotomy
  2. prone to bleeding
  3. If you are older than 80 years old
  4. In case of remote transition (M1)
  5. When long-term complications other than adjacent organ invasion (T4b) or primary tumor are needed
  6. Accompanied by intestinal obstruction, perforation, or emergency surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Operation success rate | 24hours after operation
  Surgery is complete without significant complications up to 24 hours after surgery and without conversion to other operations (laparotomy or laparoscopy)

SECONDARY OUTCOMES:
Operative outcome | immediate postoperation
  Operation time (minute)
Operative outcome | immediate postoperation
  Intraoperative bleeding volume (ml)
Operative outcome | 1 month after operation
  Length of stay (day)
Operative outcome | 1 month after operation
  Complication rate (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menon M, Shrivastava A, Tewari A, Sarle R, Hemal A, Peabody JO, Vallancien G. Laparoscopic and robot assisted radical prostatectomy: establishment of a structured program and preliminary analysis of outcomes. J Urol. 2002 Sep;168(3):945-9. doi: 10.1016/S0022-5347(05)64548-X. PMID 12187196